CLINICAL TRIAL: NCT05763732
Title: Effects of Rhythmic Auditory Stimulation (RAS) on Gait in Parkinson Disease (PD) Patients With DBS
Brief Title: Effects of RAS on Gait in PD Patients With DBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00374716
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Deep brain stimulation; Rhythmic auditory stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcomes assessor will be masked to the participants' stimulation state (OFF or ON). However, they cannot be masked whether they will receive rhythmic auditory stimulation (RAS) or not (pre-RAS or post-RAS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre RAS (No Intervention): After a 10-minute washout period, participants will receive the participants' optimized stimulation.
  1. The participants will undergo assessments to measure gait parameters and patterns during stimulation ON and OFF (Pre-RAS) using the 10-meter walk (during a 2-minute walk) and MDS-UPDRS-III rating scale.
  2. Electrophysiological activity (e.g., local field potentials, LFPs) will be collected before assessments.
- During RAS (Experimental): 1. The participants will walk to the metronome beats for four minutes (2 minutes for the same beats as baseline cadence and 2 minutes for 10% faster than baseline cadence) (RAS), and the participants' gait parameters will be recorded.
  2. Electrophysiological activity (e.g., local field potentials, LFPs) will be collected.
  Interventions: Behavioral: Rhythmic Auditory Stimulation (RAS)
- Post RAS (No Intervention): The same assessment as the Pre-RAS will be conducted (Post-RAS).

INTERVENTIONS:
Behavioral: Rhythmic Auditory Stimulation (RAS) — Rhythmic auditory stimulus (RAS) is a Neurologic Music Therapy (NMT) technique that utilizes an auditory rhythmic cue to entrain gait to a specific rhythm.
  RAS, as an anticipatory time cue, can be used as both an immediate entrainment stimulus, providing rhythmic cues during movement, and as a facilitating stimulus for planning and executing a movement to achieve more functional gait patterns. Cadence, gait velocity, and stride length are the commonly used parameters to monitor changes in a patient's gait.
  Arms: During RAS

SUMMARY:
Participants will be asked to walk along with the metronome beats (RAS) during the participants' stimulation state (ON or OFF) for four minutes for each state.

The researcher will collect the gait parameters (cadence, velocity, and stride length) of patients before, during, and after RAS in both DBS ON and OFF states.

Using MDS-UPDRS, participants' gait patterns will be collected before and after RAS while both DBS is ON and OFF. Electrophysiological activity (local field potentials, LFPs) will be collected across all stages (pre, during, and post-RAS) of evaluation.

DETAILED DESCRIPTION:
Given the evidence that rhythmic auditory stimulation (RAS) can modulate beta oscillation and improve gait parameters, the purpose of this study is to examine behavioral and neurophysiological rhythmic entrainment mechanisms.

Participants who complete the consent and enrollment process will remain for an additional up to 1 hour following the participants' routine clinic visit at the Jons Hopkins Outpatient Clinic.

The protocol will consist of two parts (DBS ON and DBS OFF). The order of stimulation states will be randomly assigned to the participants.

During DBS ON, participants will receive the participants' previously optimized stimulation after a 10-minute washout period. The researchers will measure participants' gait parameters (cadence, velocity, and stride length) with a 2-minute walk (a set distance of 10 meters during the 2-minute walk) and gait patterns using relevant items from the MDS-UPDRS-III rating scale during stimulation ON (Pre-RAS).

The participants will then walk to the metronome beats for a total of four minutes (2 minutes for the same beat as baseline cadence and 2 minutes for 10% faster than baseline cadence) (RAS), and the gait parameters will be recorded. The order of the tempo will be randomized across the participants.

Finally, after this 4-minute walk, the same assessment as for Pre-RAS will be conducted (Post-RAS).

Electrophysiological activity (local field potentials, LFPs) will be collected across all stages (pre, during, and post-RAS) of evaluation.

In DBS OFF, there will be a separate 10-minute washout period if it is taking place after DBS ON so that the participant's brain circuits can adjust to not being stimulated. Except for the DBS stimulation state, DBS OFF will follow the same protocol as DBS ON above.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson disease (PD) (and)
* PD patients who implanted Deep Brain Stimulation (DBS) of the subthalamic nucleus (STN) with PerceptTM PC

Exclusion Criteria:

* Inability or unwillingness to follow directions for study procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in gait cadence (steps/minute) | 0 minute (Baseline 1, DBS ON), 5 minutes, 10 minutes, 20 minutes (Baseline 2, DBS OFF), 25 minutes, and 30 minutes
  Gait cadence will be calculated with a 10-meter walk.
  Cadence (steps/min) = 60 / time (seconds) x # of steps
Change in gait velocity (meter/minute) | 0 minute (Baseline 1, DBS ON), 5 minutes, 10 minutes, 20 minutes (Baseline 2, DBS OFF), 25 minutes, and 30 minutes
  Gait velocity will be calculated with a 10-meter walk.
  Velocity(meter/min) = 60 / time (seconds) x 10 meter
Change in gait stride length (meter) | 0 minute (Baseline 1, DBS ON), 5 minutes, 10 minutes, 20 minutes (Baseline 2, DBS OFF), 25 minutes, and 30 minutes
  Gait stride length will be calculated with a 10-meter walk.
  Stride length (meter) = Velocity / Cadence x 2
Changes in MDS-UPDRS-III (section 3.9. Arising From Chair ) score | 0 minute (Baseline 1, DBS ON), 10 minutes, 20 minutes (Baseline 2, DBS OFF), 30 minutes
  0: Normal: No problems. Able to arise quickly without hesitation.
  1. Slight: Arising is slower than normal; or may need more than one attempt; or may need to move forward in the chair to arise. No need to use the arms of the chair.
  2. Mild: Pushes self up from the arms of the chair without difficulty.
  3. Moderate: Needs to push off, but tends to fall back; or may have to try more than one time using the arms of the chair, but can get up without help.
  4. Severe: Unable to arise without help.
Change in MDS-UPDRS-III (section 3.10. Gait) score | 0 minute (Baseline 1, DBS ON), 10 minutes, 20 minutes (Baseline 2, DBS OFF), 30 minutes
  0: Normal: No problems.
  1. Slight: Independent walking with minor gait impairment.
  2. Mild: Independent walking but with substantial gait impairment.
  3. Moderate: Requires an assistance device for safe walking (walking stick, walker) but not a person.
  4. Severe: Cannot walk at all or only with another person's assistance.
Change in MDS-UPDRS-III (section 3.11. Freezing of gait) score | 0 minute (Baseline 1, DBS ON), 10 minutes, 20 minutes (Baseline 2, DBS OFF), 30 minutes
  0: Normal: No freezing.
  1. Slight: Freezes on starting, turning, or walking through doorway with a single halt during any of these events, but then continues smoothly without freezing during straight walking.
  2. Mild: Freezes on starting, turning, or walking through doorway with more than one halt during any of these activities, but continues smoothly without freezing during straight walking.
  3. Moderate: Freezes once during straight walking.
  4. Severe: Freezes multiple times during straight walking.
Change in MDS-UPDRS-III (section 3.12. Postural stability) score | 0 minute (Baseline 1, DBS ON), 10 minutes, 20 minutes (Baseline 2, DBS OFF), 30 minutes
  0: Normal: No problems. Recovers with one or two steps.
  1. Slight: 3-5 steps, but subject recovers unaided.
  2. Mild: More than 5 steps, but subject recovers unaided.
  3. Moderate: Stands safely, but with absence of postural response; falls if not caught by examiner.
  4. Severe: Very unstable, tends to lose balance spontaneously or with just a gentle pull on the shoulders.
Change in MDS-UPDRS-III (section 3.13. Posture) score | 0 minute (Baseline 1, DBS ON), 10 minutes, 20 minutes (Baseline 2, DBS OFF), 30 minutes
  0: Normal: No problems.
  1. Slight: Not quite erect, but posture could be normal for older person.
  2. Mild: Definite flexion, scoliosis or leaning to one side, but patient can correct posture to normal posture when asked to do so.
  3. Moderate: Stooped posture, scoliosis or leaning to one side that cannot be corrected volitionally to a normal posture by the patient.
  4. Severe: Flexion, scoliosis or leaning with extreme abnormality of posture.

SECONDARY OUTCOMES:
Change in power spectrum density of Local Fields Potential (LFP) (micro-volts-squared per Hz) | 0 minute (Baseline 1, DBS ON), 5 minutes, 10 minutes, 20 minutes (Baseline 2, DBS OFF), 25 minutes, and 30 minutes
  Power spectrum density will show the strength of the variations (energy) as a function of frequency. In other words, it shows at which frequencies variations are strong and at which frequencies variations are weak.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Pantelyat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fujioka T, Ross B, Trainor LJ. Beta-Band Oscillations Represent Auditory Beat and Its Metrical Hierarchy in Perception and Imagery. J Neurosci. 2015 Nov 11;35(45):15187-98. doi: 10.1523/JNEUROSCI.2397-15.2015. PMID 26558788
- [Background] Naro A, Pignolo L, Sorbera C, Latella D, Billeri L, Manuli A, Portaro S, Bruschetta D, Calabro RS. A Case-Controlled Pilot Study on Rhythmic Auditory Stimulation-Assisted Gait Training and Conventional Physiotherapy in Patients With Parkinson's Disease Submitted to Deep Brain Stimulation. Front Neurol. 2020 Aug 4;11:794. doi: 10.3389/fneur.2020.00794. eCollection 2020. PMID 32849240
- [Background] Fujioka T, Trainor LJ, Large EW, Ross B. Beta and gamma rhythms in human auditory cortex during musical beat processing. Ann N Y Acad Sci. 2009 Jul;1169:89-92. doi: 10.1111/j.1749-6632.2009.04779.x. PMID 19673759
- [Background] Jimenez-Shahed J. Device profile of the percept PC deep brain stimulation system for the treatment of Parkinson's disease and related disorders. Expert Rev Med Devices. 2021 Apr;18(4):319-332. doi: 10.1080/17434440.2021.1909471. Epub 2021 Apr 5. PMID 33765395
- [Background] Gilron R, Little S, Perrone R, Wilt R, de Hemptinne C, Yaroshinsky MS, Racine CA, Wang SS, Ostrem JL, Larson PS, Wang DD, Galifianakis NB, Bledsoe IO, San Luciano M, Dawes HE, Worrell GA, Kremen V, Borton DA, Denison T, Starr PA. Long-term wireless streaming of neural recordings for circuit discovery and adaptive stimulation in individuals with Parkinson's disease. Nat Biotechnol. 2021 Sep;39(9):1078-1085. doi: 10.1038/s41587-021-00897-5. Epub 2021 May 3. PMID 33941932
- [Background] Torrecillos F, Tinkhauser G, Fischer P, Green AL, Aziz TZ, Foltynie T, Limousin P, Zrinzo L, Ashkan K, Brown P, Tan H. Modulation of Beta Bursts in the Subthalamic Nucleus Predicts Motor Performance. J Neurosci. 2018 Oct 10;38(41):8905-8917. doi: 10.1523/JNEUROSCI.1314-18.2018. Epub 2018 Sep 4. PMID 30181135